CLINICAL TRIAL: NCT05827224
Title: Air Optix Daily Wear Contact Lenses
Status: Completed | Type: Observational
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Other Study IDs: CLJ241-N001
Record Dates: First submitted 2023-04-13; First posted 2023-04-24 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Refractive Errors
Keywords: Contact Lenses
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (5):
- Air Optix Aqua Sphere: Lotrafilcon B spherical soft contact lenses worn in both eyes and removed daily for cleaning and disinfection
  Interventions: Device: Lotrafilcon B spherical soft contact lenses
- Air Optix plus HydraGlyde Sphere: Lotrafilcon B spherical soft contact lenses with comfort additive worn in both eyes and removed daily for cleaning and disinfection
  Interventions: Device: Lotrafilcon B spherical soft contact lenses with comfort additive
- Air Optix plus HydraGlyde Toric: Lotrafilcon B toric soft contact lenses with comfort additive worn in both eyes and removed daily for cleaning and disinfection
  Interventions: Device: Lotrafilcon B toric soft contact lenses with comfort additive
- Biofinity Sphere: Comfilcon A spherical soft contact lenses worn in both eyes and removed daily for cleaning and disinfection
  Interventions: Device: Comfilcon A spherical soft contact lenses
- Biofinity Toric: Comfilcon A toric soft contact lenses worn in both eyes and removed daily for cleaning and disinfection
  Interventions: Device: Comfilcon A toric soft contact lenses

INTERVENTIONS:
Device: Lotrafilcon B spherical soft contact lenses — Commercially available silicone hydrogel contact lenses
  Other Names: Air Optix® Aqua Sphere
  Groups: Air Optix Aqua Sphere
Device: Lotrafilcon B spherical soft contact lenses with comfort additive — Commercially available silicone hydrogel contact lenses
  Other Names: Air Optix® plus HydraGlyde® Sphere
  Groups: Air Optix plus HydraGlyde Sphere
Device: Lotrafilcon B toric soft contact lenses with comfort additive — Commercially available silicone hydrogel contact lenses
  Other Names: Air Optix® plus HydraGlyde® Toric
  Groups: Air Optix plus HydraGlyde Toric
Device: Comfilcon A spherical soft contact lenses — Commercially available silicone hydrogel contact lenses
  Other Names: Biofinity Sphere
  Groups: Biofinity Sphere
Device: Comfilcon A toric soft contact lenses — Commercially available silicone hydrogel contact lenses
  Other Names: Biofinity Toric
  Groups: Biofinity Toric

SUMMARY:
The purpose of this Post-Market Clinical Follow-Up (PMCF) study is to assess long term performance and safety of Air Optix Aqua, Air Optix plus HydraGlyde Sphere, and Air Optix plus HydraGlyde Toric soft contact lenses in a real-world setting when worn as daily wear.

DETAILED DESCRIPTION:
This is a non-interventional/observational study designed as a retrospective chart review. Study sites will identify charts within their existing databases in a fair and consistent manner, e.g., reviewing all eligible charts in reverse chronological order by year of baseline visit. The baseline visit will be defined as the first office visit where an eye care practitioner provided an in-person office biomicroscopy exam to the patient, before or during which a contact lens prescription for the study or comparator contact lenses was released. Subjects meeting the eligibility criteria will be enrolled in the study.

ELIGIBILITY:
Key Inclusion Criteria:

* Manifest refraction cylinder less than or equal to 0.75 diopter (D) in each eye at baseline (sphere wearers only);
* Best corrected visual acuity (BCVA) of 20/25 Snellen or better in each eye at baseline;
* Must have worn or be wearing Air Optix Aqua Sphere, Air Optix plus HydraGlyde Sphere, Air Optix plus HydraGlyde Toric, Biofinity Sphere or Biofinity Toric for at least 1 year in a daily wear modality, as determined by the Investigator;
* Other protocol-defined inclusion criteria may apply.

Key Exclusion Criteria:

* Have worn or be wearing Air Optix Aqua Sphere, Air Optix plus HydraGlyde Sphere, Air Optix plus HydraGlyde Toric, Biofinity Sphere, or Biofinity Toric contact lenses in an extended wear modality;
* Any recurrent history or active anterior segment infection, inflammation or abnormality contraindicating regular contact lens wear at baseline;
* Use of systemic or ocular medications contraindicating regular contact lens wear at baseline and/or during the period of the retrospective chart collection;
* Slit lamp findings, including signs of pathological dry eye, that would contraindicate regular contact lens wear;
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Investigators will enroll charts following a pre-identified process.
Sampling Method: Non-Probability Sample
Enrollment: 312 (Actual)
Dates: Start 2023-08-02 (Actual); Primary Completion 2024-07-17 (Actual); Study Completion 2024-07-17 (Actual)

PRIMARY OUTCOMES:
Distance visual acuity (VA) with study lenses | Up to Year 1
  The subject's chart will be reviewed for distance visual acuity at baseline and at 1 year following the baseline exam.
Incidence of corneal infiltrative events | Up to Year 1
  The subject's chart will be reviewed for incidences of corneal infiltrative events occurring after the baseline exam.
Incidence of microbial keratitis | Up to Year 1
  The subject's chart will be reviewed for incidences of microbial keratitis occurring after the baseline exam.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Lead, Vision Care, Study Director — Alcon Research, LLC
Locations (5):
- United States (5):
  - Vision Health Institute, Orlando, Florida
  - Complete Eye Care of Medina, Medina, Minnesota
  - Koetting Associates, St Louis, Missouri
  - Toyos Clinic, Nashville, Tennessee
  - Smith Bowman Ophthalmology, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No